CLINICAL TRIAL: NCT02286505
Title: Automated Brain Morphometry for Dementia Diagnosis
Acronym: BrainMeasure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Collaborators: Imperial College London (Other); University of Sussex (Other); IXICO Limited (Unknown); Cambridge Cognition Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 101353
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brain Morphometry (Experimental): Quantitative, automated reading of hippocampal volume from MRI scans, complemented by a general measure of brain atrophy, in addition to standard neuroradiological report.
  Interventions: Device: Brain Morphometry; Other: Standard radiological assessment
- Standard radiological assessment. (Other): Standard neuroradiological report of the structural MRI only.
  Interventions: Other: Standard radiological assessment

INTERVENTIONS:
Device: Brain Morphometry — Quantitative, automated reading of hippocampal volume from MRI scans, complemented by a general measure of brain atrophy, in addition to standard neuroradiological report.
  Arms: Brain Morphometry
Other: Standard radiological assessment — Standard neuroradiological report produced by qualitative examination of structural MRI scan by trained neuroradiologist.

SUMMARY:
Early dementia diagnosis improves patient and carer experience, links them to appropriate care and support and enables timely symptomatic treatment. The guidelines of the UK National Institute for Health and Care Excellence recommend brain Magnetic resonance imaging (MRI) to assist with the diagnosis in suspected dementia. Recently, computerised analysis of MRI scans, also known as automated brain morphometry, has shown potential to detect the brain changes characteristic of early dementia, and may therefore be a useful addition to the standard reporting performed by a neuroradiologist. The present pilot study will assess whether adding brain morphometric analysis to the usual diagnostic pathway improve diagnosis in clinical practice as an addition to the existing diagnostic pathway in a memory clinic setting. The main purpose of the study is to compare measures of the clinicians diagnostic confidence in patients with and without brain morphometry.

ELIGIBILITY:
Inclusion Criteria:

* Subjects referred to a South London and Maudsley (SLaM) memory clinic for suspected dementia.
* Cognitive scores (standardised MMSE of 15 or more inclusive) and impairment in activities of daily living consistent with a diagnosis of mild to moderate dementia or mild cognitive impairment.
* Working knowledge of English.
* Must consent to the imaging and follow-up aspects of the study. If the patient lacks capacity to consent to the study, they will not be invited to participate.
* If the patient has a partner or carer able to provide an independent evaluation of functioning and able and willing to be involved in a follow-up interview about their experience of the diagnostic process, the carer should also consent to participate in the study.

Exclusion Criteria:

* Contraindications for MRI
* Patients 50 or younger (cognitive impairment in this younger population is only exceptionally due to a neurodegenerative condition). There are no upper age limits.

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Difference in confidence in the clinical diagnosis | 12 weeks
  Difference in confidence of the clinical diagnosis between the two arms of the trial (patient with and without quantitative brain morphometric analysis). This is a number for each subject ranging from 1 (not at all confident) to 5 (extremely confident), as measured by a questionnaire completed by the clinician at the time of final diagnosis.

SECONDARY OUTCOMES:
Time to diagnosis. | 12 weeks
  Comparing time from referral to diagnosis in patients with and without brain morphometry.

OTHER OUTCOMES:
Time to treatment | 12 weeks
  Time to prescription of symptomatic treatment (cholinesterase inhibitors or memantine) in patients with and without the brain morphometry analysis.
Patient and carer satisfaction | 12 weeks
  Satisfaction in the diagnostic process as measured by questionnaire administered at time of final diagnosis to patient and carer, if available.

CONTACTS AND LOCATIONS:
Overall Officials: Sergi Costafreda-Gonzalez, MD, PhD, Principal Investigator — King's College London; Andrew Simmons, PhD, Principal Investigator — King's College London
Locations (1):
- Old Age Psychiatry and Dementia Clinical Academic Group, South London and Maudsley NHS Foundation Trust and King's College London, London, London, United Kingdom